CLINICAL TRIAL: NCT01520441
Title: H-25362: Effect of Botulinum Neurotoxin Type A Prostate Injections on Neurogenesis and Gene Profile Expression in Men With Localized Prostate Cancer and Lower Urinary Tract Symptoms/BPH (Protocol # 05-09-30-03)
Brief Title: BOTOX in Men With Prostate Cancer With Lower Urinary Tract Symptoms(LUTS)/Benign Prostatic Hyperplasia (BPH)
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Gustavo Ayala, Professor and Distinguished Chair in Pathology and Laboratory Medicine, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-25362
Record Dates: First submitted 2012-01-24; First posted 2012-01-30 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Prostate Cancer; Benign Prostatic Hyperplasia; Enlarged Prostate With Lower Urinary Tract Symptoms (LUTS)
Keywords: Botulinum Toxin; Prostate Cancer; BPH; LUTS
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Hyperplasia | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BOTOX Injection (Experimental): A total of 200 units of BoNT-A diluted in 4ml of preservative free saline will be injected into the right prostate lobe (i.e. transition and peripheral zones). A similar injection template with 1.0ml volume injections of saline will be injected into the left prostate lobe (2 injections in transition zone, 2 injections in peripheral zone for total volume of 4ml).
  Interventions: Drug: BOTOX

INTERVENTIONS:
Drug: BOTOX — A total of 200 units of BoNT-A diluted in 4ml of preservative free saline will be injected into the right prostate lobe (i.e. transition and peripheral zones). A similar injection template with 1.0ml volume injections of saline will be injected into the left prostate lobe (2 injections in transition zone, 2 injections in peripheral zone for total volume of 4ml).
  Other Names: onabotulinumtoxinA

SUMMARY:
This is a pilot study examining biological endpoints in men with localized prostate cancer who are scheduled to have radical prostatectomies and men with Benign Prostatic Hyperplasia/Lower Urinary Tract Symptoms (BPH/LUTS) following botulinum toxin type A (BoNT-A) injection. Patients will serve as their own controls by receiving BoNT-A injections into the right peripheral and transition zones and sham saline injections into the left peripheral and transition zones.

DETAILED DESCRIPTION:
For the purposes of this study, patients are treated with the presentation of botulinum toxin type A which is marketed in the U.S. as BOTOX® by Allergan. BOTOX® is a purified neurotoxin complex supplied as a sterile, vacuum dried purified botulinum toxin type A, produced from fermentation of Clostridium botulinum type A.

A primary aim of this study is to determine the molecular effects of BoNT-A injection on human BPH tissues. While the majority of BoNT-A injections in humans target BPH in the transition zone, innervation is most abundant in the peripheral zone of the prostate where the majority of prostate cancers develop. In fact, recent studies have demonstrated the importance of neurogenesis and axogenesis in the spread of human prostate cancer. In addition, in vitro studies have shown that BoNT-A has antiproliferative effects on human prostate cancer cell lines.

Thus, a second aim of this proposal is to determine profile changes in high-grade prostatic intraepithelial neoplasia (HGPIN) and prostate cancer following BoNT-A injection into the peripheral zone. The investigators will also determine the effects of BoNT-A on the genetic profile of normal tissue. The investigators study population will be men with clinically localized prostate cancer. Men will be injected on one side in both their transition and peripheral zones with 100U BoNT-A (i.e. Botox®, Allergan, Inc.), respectively, one month prior to their scheduled radical prostatectomy. Sham saline injection of the other side of the prostate (transition and peripheral zones) will be used as an internal control. The investigators will inject the other lobe of the prostate with saline to account for any denervating effects of "wet needling." Patients will undergo radical prostatectomy without any changes to standard of care. The strategy has been used in the investigators Institution previously to determine the efficacy of gene therapy 22 and targeted drugs. However, and unlike the investigators previous neoadjuvant trials, the investigators will not power this study to look at the effects of Botox on biochemical recurrence free survival. This study only has biologic endpoints and no survival endpoints."

A third aim of the study will be to examine changes in vas deferens function following prostate treatment with BoNT-A. The investigators plan to harvest a 2.5 cm segment from the distal vas deferens on either side (i.e. Saline treated and BoNT-A treated) before entry into the prostate will be isolated and placed in oxygenated krebs solution for transport to the research laboratory.

Patients will have 3 visits to the clinic and two telephone calls during their participation in this study. The last visit is about 4 weeks after the injection.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven, clinically localized prostate cancer
* Low risk for recurrence defined as a Kattan nomogram score of less than 115, or a serum PSA < 10ng/ml, or an individual Gleason grade of 3 or lower, or clinical stage T2b or below.
* Candidates diagnosed with localized prostate cancer must have agreed to radical prostatectomy.
* Voided volume greater than or equal to 125 ml.
* Maximum urinary flow less than 15 ml/sec.
* American Urological Association (AUA) symptom severity score greater than or equal to 8.
* Patient signed informed consent prior to the performance of any study procedures.
* Patient able to complete the study protocol in the opinion of the investigator.

Exclusion Criteria:

* Any prior surgical intervention for BPH.
* Current diagnosis of acute or chronic prostatitis (which may cause LUTS that mimic BPH).
* History of bladder stones.
* Overactive bladder without bladder outlet obstruction.
* Enrolled in another treatment trial for any disease within the past 30 days.
* Previous exposure to botulinum toxin.
* Post void residual greater than 350 ml.
* Clinically significant renal or hepatic impairment as determined by abnormal creatinine or AST levels (based on local institutional values).
* Daily use of a pad or device for incontinence required.
* Episode of unstable angina pectoris, myocardial infarction, transient ischemic attack, or cerebrovascular accident (stroke) within the past 6 months.
* On aminoglycosides or any drug that interfere with neuromuscular transmission.
* Eaton-Lambert syndrome, hemophilia, hereditary clotting factors deficiency, or bleeding diathesis.
* Penile prosthesis or artificial urinary sphincter.
* History or current evidence of carcinoma of the bladder; pelvic radiation, hormonal treatment or surgery; urethral stricture; or bladder neck obstruction.
* Known primary neurologic conditions such as multiple sclerosis, myasthenia gravis or Parkinson's disease, or other neurological diseases known to affect bladder function.
* Two documented urinary tract infections of any type in the past year (UTI defined as greater than 100,000 colonies per ml urine from midstream clean catch or catheterized specimen).
* Patients must be off aspirin, non-steroidal anti-inflammatory drugs (NSAIDS), and Coumadin for 7 or more days prior to botulinum toxin injection.
* Any serious medical condition likely to impede successful completion of the study, such as certain mental disorders, hypersensitivity to botulinum toxin or anesthetics used in the study, syncope, uncontrolled diabetes.
* Patients will be excluded if they have depressed hematopoietic functions (platelet count <100,000/cm3, hemoglobin <8,5 mg/dl; absolute neutrophil count <1000/cm3).

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Determination the effects of BoNT-A injection on BPH and prostate cancer tissues. | 3 years
  The prostate tissue taken from each lobe will be compared to determine if the injection of BOTOX has effected the genetic profile.

SECONDARY OUTCOMES:
Determination of BOTOX prostate injection on vas deferens tissue | 3 years
  Any changes to the vas deferens tissue after BOTOX injection, will be noted.

CONTACTS AND LOCATIONS:
Overall Officials: Gusatavo E. Ayala, MD, Principal Investigator — University of Texas Houston Health Science Center
Locations (1):
- University of Texas Houston - Medical School, Houston, Texas, United States

REFERENCES:
- [Background] Chancellor MB, Smith CP: Botulinum Toxin in Urology. First Edition. New York: Springer, Aug 2011. (Book)
- [Background] Smith CP. Botulinum toxin in the treatment of OAB, BPH, and IC. Toxicon. 2009 Oct;54(5):639-46. doi: 10.1016/j.toxicon.2009.02.021. Epub 2009 Mar 4. PMID 19268490
- [Background] Crawford ED, Hirst K, Kusek JW, Donnell RF, Kaplan SA, McVary KT, Mynderse LA, Roehrborn CG, Smith CP, Bruskewitz R. Effects of 100 and 300 units of onabotulinum toxin A on lower urinary tract symptoms of benign prostatic hyperplasia: a phase II randomized clinical trial. J Urol. 2011 Sep;186(3):965-70. doi: 10.1016/j.juro.2011.04.062. Epub 2011 Jul 24. PMID 21791356